CLINICAL TRIAL: NCT03112109
Title: SmartCare Project: Joining up ICT and Service Processes for Quality Integrated Care in Europe
Brief Title: SMARTCARE Project: Deploying Integrated Health & Social Services for Independent Living by Older People
Acronym: SmartCare
Status: Completed | Type: Observational
Sponsor: Him SA (Other)
Responsible Party: Sponsor
Other Study IDs: SmartCare_EC_Grant_No.325158
Record Dates: First submitted 2017-03-08; First posted 2017-04-13 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Frail Elderly Syndrome; Congestive Heart Failure; Falls Prevention
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: Patients receiving 'new care'
  Interventions: Other: 'New care'
- Control group: Patients receiving 'old / usual care'

INTERVENTIONS:
Other: 'New care' — Frail elderly receiving care within new organisational models delivering integrated healthcare (IHC) supported by ICT infrastructure (electronically shared-care platform) as provided by pilot sites individually.
  Groups: Intervention Group

SUMMARY:
Against the background of the European Innovation Partnership on Active & Healthy Ageing, SmartCare aims to define a common set of standard functional specifications for an open ICT platform enabling the delivery of integrated care to older European citizens.

In the context of SmartCare, a total of 23 regions and their key stakeholders will define a comprehensive set of integration building blocks around the challenges of data-sharing, coordination and communication. Nine regions will then deploy integrated health & social services to combat a range of threats to independent living commonly faced by older people, while the others will prepare for early adoption, possibly in the framework of new ICT PSP projects. In a rigorous evaluation approach, the deployment sites will produce and document much needed evidence on the impact of integrated care, developing a common framework suitable for other regions in Europe. The organisational and legal ramifications of integrated care will be analysed to support long term sustainability and upscaling of the services.

SmartCare services will provide full support to cooperative delivery of care, integrated with self-care and across organisational silos, including essential coordination tools such as shared data access, care pathway design and execution, as well as real time communication support to care teams and multi-organisation access to home platforms. In addition, they will empower all older people according to their mental faculties to take part in effective management of their health, wellness, and chronic conditions, and maintain their independence despite increasing frailty.

The SmartCare services build on advanced ICT already deployed in the pioneer regions, including high penetrations of telecare and telemonitoring home platforms. In SmartCare, these platforms are to be opened to cross-sectorial care teams, improving the ability of older people to better manage their chronic conditions at home and deal with their increasing frailty. System integration will be based, whenever possible, on open standards' multivendor interoperability will be strongly encouraged.

DETAILED DESCRIPTION:
This trial will evaluate the functions and impacts of the SmartCare pilot services from the point of view of the different principal roles/stakeholders, such as end users (care recipients), voluntary and non-voluntary informal carers, formal care staff/professionals, managers and fund-holders. Evaluation of integrated care service delivery processes (process evaluation) will improve the current scientifically based knowledge base on barriers and facilitators towards integrated care delivery.

Comparators were chosen to be current delivery of health and social care processes ('normal care'), as provided by pilot sites individually. The project uses local scenarios as the comparator in order to enable the evidence generated to contribute to local decision making on using the technologies. Thus, the control groups were as similar as possible to the intervention groups (receiving 'new care'). In addition, a number of possible confounding factors were measured for all participants.

The overall aim of the scientific studies carried out in SmartCare is: To identify the differences induced by implementing ICT supported integrated health and social care.

Any impact that ICT supported integrated health and social care might have on all users will be the subject of analyses according to the framework presented in the MAST model (Kidholm et al. 2012).

In addition, the objectives that will be tested in SmartCare are:

* Difference in number of contacts to health care.
* Difference in number of contacts to social care.
* Differences in use of health care services.
* Differences in use of social care services.
* Differences in costs.
* Differences in organisational aspects caused by implementing ICT supported integrated care.
* Difference in end-user empowerment.
* Difference in end-user satisfaction.

ELIGIBILITY:
Inclusion criteria for end users:

* Provided with both health and social care.
* Congestive heart failure: for RSD pilot site.
* Frail elderly: for Aragon pilot site.

Exclusion criteria for end users:

* No exclusion criteria.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Interventions will be provided by a combination of health care, social care, volunteer sector care providers, and informal carers to the population samples to be drawn either by randomisation or consecutive inclusion of either intervention or control end-users determined by geographical areas (pilot sites). Additionally, these inclusion criteria for end users are applicable:
  Thus, the professionals that are involved in providing any type of health and/or social care for the included citizens will be enrolled as intervention performers and as users of the interventions.
Sampling Method: Probability Sample
Enrollment: 2111 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Change in services consumption | Healthcare services consumption measured at individual level, per individual client / citizen / carer, based on differences ('change') between measurements at (a) baseline (month 0), (b) midterm (12 months) and (c) end (24 months) of study
  Change in healthcare and social care services consumption measured based on total count of healthcare services consumption, measured based on total count of number of contacts with healthcare services/professionals

SECONDARY OUTCOMES:
Blood pressure | Blood pressure measured in mmHG, at individual level, per individual client / citizen at baseline, midterm (12 months) and end (24 months) of study
  Blood pressure as part of disease specific health status measurements
Blood glucose | Blood glucose measured in mg/dl, at individual level, per individual client / citizen / carer at baseline, midterm (12 months) and end (24 months) of study
  Blood glucose as part of disease specific health status measurements
Cholesterol | Cholesterol measured in mmol/ltr, at individual level, per individual client / citizen at baseline, midterm (12 months) and end (24 months) of study
  Cholesterol as part of disease specific health status measurements
General health and wellbeing / Indicator for health status | General health and wellbeing (SF 36 v2) measured with questionnaire, at individual level, per individual client / citizen at baseline and end (24 months) of study
  General health and wellbeing based on v2 of the SF 36 questionnaire
Indicator for health status: Barthel | Indicator for health status as measured with Barthel Index measured with questionnaire, at individual level, per individual client / citizen at baseline and end (24 months) of study
  Indicator for health status as measured with Barthel Index
Indicator for health status: Timed up & go | Indicator for health status measured with Timed up and Go test, at individual level, per individual client / citizen at baseline and end (24 months) of study
  Indicator for health status as measured with Timed up and Go test
Quality of Life of family carers: CASP | Quality of Life of family carers measured with CASP-19, at individual level, per carer at baseline and end (24 months) of study
  Quality of Life of family carers, based on levels of Control, Autonomy, Pleasure and Self-realization (with CASP-19 questionnaire)
Anxiety and depression | Anxiety and depression levels in end users Quality of Life of family carers measured with HADS Scale, at individual level, per citizen / client at baseline and end (24 months) of study
  Anxiety and depression according as part of psychological status, based on HADS scale
Depression in elderly | Depression in elderly in end users measured with (GDS-15), at individual level, per citizen / client at baseline and end (24 months) of study
  Depression in elderly as part of psychological status, based on Geriatric Depression Scale-15 (GDS-15)
Isolation | Level of isolation in elderly in end users measured with Perceived Isolation Questionnaire, at individual level, per citizen / client at baseline and end (24 months) of study
  Level of isolation according to Perceived Isolation Questionnaire as part of psychological status
Carer burden | Level of carer burden measured with ZBI in carers measured at individual level, per caregivers at baseline and end (24 months) of study
  Level carer burden according to Zarit Burden Interview (ZBI) as part of psychological status
Carer difficulties, satisfaction and management in caring - I | Level of carer difficulties, satisfaction and management in caring measured with CADI in carers measured at individual level, per caregivers at baseline and end (24 months) of study
  Level of carer difficulties, satisfaction and management in caring according to: Carer Assessment of Difficulty Index (CADI)
Carer difficulties, satisfaction and management in caring - II | Level of carer difficulties, satisfaction and management in caring measured with CASI suite in carers measured at individual level, per caregivers at baseline and end (24 months) of study
  Level of carer difficulties, satisfaction and management in caring according to Carer Assessment of Satisfaction Index (CASI)
Carer difficulties, satisfaction and management in caring - III | Level of carer difficulties, satisfaction and management in caring measured with CAMI suite in carers measured at individual level, per caregivers at baseline and end (24 months) of study
  Level of carer difficulties, satisfaction and management in caring according to: Carer Assessment of Management Index (CAMI) as part of psychological status
Death | Death as adverse outcome measure as registered at end of study (24 months)
  Death as adverse outcome measure

IPD SHARING:
Plan to Share IPD: No